CLINICAL TRIAL: NCT01190761
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Galantamine 4 mg Tablet and Reminyl Following a 4 mg Dose in Healthy Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Galantamine 4 mg Tablet and Reminyl Following a 4 mg Dose in Healthy Subjects Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 40464
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Galantamine; Reminyl; Galantamine hydrobromide; Healthy subjects
MeSH Terms: interventions — Galantamine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Galantamine 4 mg Tablet, single dose
  Interventions: Drug: Galantamine 4 mg Tablet, single dose
- B (Active Comparator): Reminyl 4 mg Tablet, single dose
  Interventions: Drug: Reminyl 4 mg Tablet, single dose

INTERVENTIONS:
Drug: Galantamine 4 mg Tablet, single dose — A: Experimental Subjects received Purepac Pharmaceutical, Company, U.S.A. formulated products under fed conditions
  Other Names: Galantamine
  Arms: A
Drug: Reminyl 4 mg Tablet, single dose — B: Active comparator Subjects received Janssen Pharmaceutica Products,U.S.A., formulated products under fed conditions
  Other Names: Galantamine hydrobromide
  Arms: B

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of Purepac, a subsidiary of Alpharma Inc., U.S.A., galantamine and Janssen Pharmaceutica Products, L.P., U.S.A. (Reminyl),galantamine, administered as a 1 x 4 mg tablet, under fed conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, 2-period, 2-sequence, crossover design.

Official Title: Randomized, 2-Way Crossover, Bioequivalence Study of Galantamine 4 mg Tablet and Reminyl Following a 4 mg Dose in Healthy Subjects Under Fed Conditions.

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may use various media types (e.g. radio, newspaper, SFBC Anapharm Web site, SFBC Anapharm volunteers' database). Subjects must meet all of the following criteria in order to be included in the study:

* Male or female, smoker or non-smoker, 18 years of age and older
* Capable of consent.
* BMI2:19.0 and <30.0 kg/rn".

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

• Clinically significant illnesses within 4 weeks prior to the administration of the study medication.

Clinically significant surgery within 4 weeks prior to the administration of the study medication.

* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HN at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
* Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to heparin, galantamine, other tertiary alkaloid derivatives or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoine, glucocorticoids, omeprazole; examples of inhibitors: antidepressant (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion ofthe drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary (including asthma and COPD), hematologic, immunologic, psychiatric, or metabolic disease.

Use of prescription medication (including hormone therapy) within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption or hormonal contraceptive.

* Difficulty to swallow study medication.
* Smoking more than 25 cigarettes per day.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug (other than hormonal contraceptive) within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days,
* 301 mL to 500 mL of whole blood within 45 days, or
* more than 500 mL of whole blood within 56 days prior to drug administration.
* History of "sick sinus syndrome" or other supraventricular cardiac conduction disorders,active coronary artery disease or congestive heart failure.
* History of unexplained syncopal episodes.
* Consumption of food or beverages containing grapefruit (e.g. fresh, canned, or frozen)within 7 days prior to administration of the study medication.
* History of ulcer disease.
* History of asthma or obstructive pulmonary disease.
* History of seizure disorder.
* Breast-feeding.
* Positive urine pregnancy test at screening.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. Acceptable methods of contraception:
* condom + spermicide;
* diaphragm + spermicide;
* intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration);
* hormonal contraceptives (starting at least 4 weeks prior to study drug administration).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-12; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D., Principal Investigator — SFBC Anapharm
Locations (1):
- SFBC Anapharm, Sainte-Foy, Quebec, Canada